CLINICAL TRIAL: NCT00002665
Title: TREATMENT OF ADULT ACUTE LYMPHOBLASTIC LEUKEMIA: PHASE II TRIALS OF AN INDUCTION REGIMEN INCLUDING PEG-L-ASPARAGINASE, WITH OR WITHOUT PIXY, IN PREVIOUSLY UNTREATED PATIENTS, FOLLOWED BY ALLOGENEIC BONE MARROW TRANSPLANTATION OR FURTHER CHEMOTHERAPY IN FIRST COMPLETE REMISSION
Brief Title: SWOG-9400 Combination Chemotherapy With or Without Bone Marrow Transplantation in Treating Patients With Previously Untreated Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWOG-9400; SWOG-9400 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia; Neutropenia; Thrombocytopenia
Keywords: untreated adult acute lymphoblastic leukemia; L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; neutropenia; thrombocytopenia
MeSH Terms: conditions — Leukemia; Neutropenia; Thrombocytopenia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Etoposide; Leucovorin; Mercaptopurine; Methotrexate; Prednisone; Thioguanine; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: asparaginase — 10,000 units/d IV or IM 15 - 24
Drug: cyclophosphamide — con: 650 mg/m2 IV 1, 15, 29 maint: 650 mg/m2 IV 1
Drug: cytarabine — cons: 75 mg/m2/d IV Push 2 - 5, 9 - 12, 6 - 19, 23 - 26
Drug: daunorubicin hydrochloride — ind: 60 mg/m2 IV 22 and 23
Drug: dexamethasone — main: 10 mg/m2/day PO 1 - 28
Drug: doxorubicin hydrochloride — main: 25 mg/m2 IV 1, 8, 15, and 22
Drug: etoposide — 60 mg/kg based on ideal body weight day -3
Drug: leucovorin calcium — 5 mg q 6 hours for 4 doses, PO 1, 3, 8, 11 after each methotrexate if WBC < 3,000 /μl
Drug: mercaptopurine — con: 60 mg/m2 PO 1 - 28
Drug: methotrexate — 10 mg/m2 IT or IV, d 2, 9, 16, and 23; Maximum 15 mg/admin
Drug: prednisone — ind: 60 mg/m2/d PO 1 - 21*, 22 - 28 Patients will receive full dose through day 8 and then tapered to zero between Day 29 and 42.
  ind2: 60 mg/m2/d PO through day 42
Drug: thioguanine — main: 60 mg/m2/day PO 1 - 14
Drug: vincristine sulfate — ind: 1.4 mg/m2 2 mg max, IV 1, 8, 15, and 22 ind2: 1.4 mg/m2 2 mg max IV 29 and 36 main: 1.5 mg/m2 2 mg max, IV 1, 8, 15, and 22
Procedure: allogeneic bone marrow transplantation — day 0
Radiation: radiation therapy — day -7 through day -4 total dose of radiation is 1,320 cGy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with or without bone marrow transplantation in treating patients who have acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate if front line induction therapy with daunorubicin, vincristine, prednisone, and asparaginase is sufficiently effective to warrant a phase III trial in patients with acute lymphocytic leukemia (ALL). II. Assess the toxicity of this regimen in this patient population. III. Assess disease free and overall survival and toxicity associated with allogeneic bone marrow transplantation for ALL patients in first remission following induction and consolidation therapy. IV. Assess disease free and overall survival and toxicity associated with sequential regimens of mercaptopurine, methotrexate and vincristine, doxorubicin, dexamethasone, and cyclophosphamide, thioguanine, and cytarabine in ALL patients in first remission who are ineligible for allogeneic bone marrow transplantation. V. Evaluate the prognostic significance of cell surface immunophenotype, Philadelphia chromosome, and polymerase chain reaction detected BCR/abl fusion in this patient population.

OUTLINE: Patients are stratified according to age (15 to 29 vs 30 to 49 vs 50 to 65), performance status (0-1 vs 2-3), participating center, and candidate for allogeneic bone marrow transplantation (yes vs no). Patients receive induction chemotherapy consisting of daunorubicin IV on days 1-3, vincristine IV on days 1, 8, 15, and 22, oral prednisone on days 1-28, and asparaginase IV or intramuscularly (IM) on days 15-24. Patients with persistent leukemia on day 21, receive additional induction therapy consisting of daunorubicin IV on days 22 and 23, vincristine IV on days 29 and 36, and oral prednisone continuing to day 42. Patients with CNS leukemia receive additional therapy beginning on day 1 of induction chemotherapy consisting of methotrexate intrathecally (IT) or intraventricularly twice weekly until blasts are absent in spinal fluid. Patients receive oral leucovorin calcium every 6 hours for a total of 4 doses following each IT dose in the absence of blood count recovery. Following absence of spinal fluid blasts, patients receive methotrexate IT or intraventricularly weekly for 4 weeks then monthly for 1 year. Patients also receive cranial radiotherapy during consolidation therapy 5 days a week for 2.5 weeks. Patients with A1 bone marrow receive consolidation therapy following completion of induction therapy and blood count recovery. Patients receive consolidation therapy consisting of cyclophosphamide IV on days 1, 15, and 29, cytarabine IV on days 2-5, 9-12, 16-19, and 23-26, oral mercaptopurine on days 1-28, and methotrexate IT on days 2, 9, 16, and 23. Following completion of consolidation therapy, patients eligible for allogeneic bone marrow transplantation receive total body radiotherapy 3 times a day on days -7, -6, -5, and twice on day -4, and eptoposide IV over 4 hours on day -3. Patients undergo allogeneic bone marrow transplantation on day 0. Following completion of consolidation therapy, patients ineligible for allogeneic bone marrow transplantation receive maintenance therapy consisting of oral mercaptopurine on days 1-63, and oral methotrexate on days 1, 8, 15, 22, 29, 36, 43, 50, and 57. Patients receive subsequent courses of maintenance therapy when blood counts recover. Patients receive a second course of maintenance therapy consisting of vincristine IV on days 1, 8, 15, and 22, doxorubicin IV on days 1, 8, 15, and 22, and oral dexamethasone on days 1-28. Patients receive a third course consisting of cyclophosphamide IV on day 1, oral thioguanine on days 1-14, and cytarabine IV on days 3-6 and 10-13. Patients receive a fourth course consisting of oral mercaptopurine and oral methotrexate daily for 2 years. Patients are followed monthly for 6 months and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 25-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed acute lymphocytic leukemia FAB class L1-L2 Mixed immunophenotypic markers with no cytochemical myeloid markers allowed No non-Hodgkin's lymphoma No chronic myelogenous leukemia in blast crisis Concurrent registration on the cytogenetics protocol SWOG-9007 required

PATIENT CHARACTERISTICS: Age: 15 to 65 Performance status: SWOG 0-3 Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2 times normal (unless elevation due to leukemia) AST no greater than 3 times normal (unless elevation due to leukemia) No chronic liver disease Renal: Creatinine no greater than 2 times normal Cardiovascular: Left ventricular ejection fraction at least 50% by MUGA or echocardiogram No symptomatic congestive heart failure No symptomatic coronary artery disease No cardiomyopathy No uncontrolled arrhythmia Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: No prior remission induction chemotherapy for acute lymphocytic leukemia

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1995-07; Primary Completion 2001-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
response

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Forman, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (83):
- United States (83):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Pullarkat V, Slovak ML, Kopecky KJ, Forman SJ, Appelbaum FR. Impact of cytogenetics on the outcome of adult acute lymphoblastic leukemia: results of Southwest Oncology Group 9400 study. Blood. 2008 Mar 1;111(5):2563-72. doi: 10.1182/blood-2007-10-116186. Epub 2007 Dec 21. PMID 18156492
- [Result] Sala-Torra O, Gundacker HM, Stirewalt DL, Ladne PA, Pogosova-Agadjanyan EL, Slovak ML, Willman CL, Heimfeld S, Boldt DH, Radich JP. Connective tissue growth factor (CTGF) expression and outcome in adult patients with acute lymphoblastic leukemia. Blood. 2007 Apr 1;109(7):3080-3. doi: 10.1182/blood-2006-06-031096. PMID 17170128
- [Result] Sala-Torra O, Gundacker HM, Stirewalt DL, et al.: CTGF (CCN2) predicts OS and DFS in adult acute lymphoblastic leukemia. [Abstract] Blood 106 (11): A-336, 2005.
- [Result] Slovak ML, Kopecky KJ, Gundacker H, et al.: Clinical significance of cytogenetic abnormalities in adult acute lymphoblastic leukemia (ALL): a Southwest Oncology Group (SWOG) study (S9400). [Abstract] Blood 102 (11 Pt 1): A-2223, 2003.
- [Result] Boldt DH, Gundacker HM, Lee DY, et al.: Analysis of multidrug resistance gene-1 (MDR1) expression and function in adult acute lymphoblastic leukemia (ALL). A Southwest Oncology Group (SWOG) study. [Abstract] Blood 100 (11 Pt 1): A-2991, 2002.
- [Result] Gazitt Y, Lee D, Wang ME, et al.: Functional MDR1 expression in adult acute lymphoblastic leukemia (ALL). Blood 92 (10 Suppl 1): A-2788, 676a, 1998.